CLINICAL TRIAL: NCT03968107
Title: Diagnostic Performance of Antenatal Ultrasound in the Localization of Intestinal Structures Involved in Malrotation With a Higher-risk of Volvulus
Brief Title: Diagnostic Performance of Antenatal Ultrasound for High-Risk Intestinal Malrotation
Acronym: MALGRE
Status: Terminated | Type: Observational
Why Stopped: The study was terminated prematurely, as the inclusion period ended on 11/27/2024. Of the 103 patients planned, 77 were included.
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0454 UF 7722; 2019-A00614-53 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related
Keywords: malrotation; intestinal structures; mesenteric vessels; prenatal diagnosis; congenital abnormalities; digestive system abnormalities; torsion abnormality; intestinal volvulus
MeSH Terms: conditions — Volvulus Of Midgut; Congenital Abnormalities; Digestive System Abnormalities; Torsion Abnormality; Intestinal Volvulus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with a pregnancy of at least 31 weeks: All pregnant women with a pregnancy of at least 31 weeks and having to perform a fetal MRI to identify a cerebral, pulmonary or renal fetal malformation, or due to a diagnostic doubt on ultrasound on an abnormality of these structures, will be proposed inclusion in the study.
  Interventions: Other: Reference ultrasound examination

INTERVENTIONS:
Other: Reference ultrasound examination — Use of antenatal ultrasound examination to visualize and position the intestinal structures involved in digestive malrotation at high risk of volvulus and comparison to fetal MRI results.
  Other Names: Fetal MRI; Comparison of both results

SUMMARY:
The aims of this study are:

* To assess the performance of third-trimester ultrasound scan in the localization of intestinal structures (small bowel, gut, mesenteric vessels..) involved in malrotations with a higher-risk of volvulus compared to a gold standard based on fetal magnetic resonance imaging (MRI).
* To describe normal meconium progression (ultrasound and MRI), prenatal anatomical variants of the fetal digestive tract, and interobserver agreement on prenatal ultrasound.

DETAILED DESCRIPTION:
Introduction: Intestinal malrotation is a rare congenital anomaly resulting from abnormal rotation and fixation of the intestine during embryonic development. It is rarely asymptomatic and most often presents in the neonatal period with obstructive complications, including duodenal obstruction and, most critically, midgut volvulus. Midgut volvulus constitutes a surgical emergency due to the risk of extensive intestinal ischemia and necrosis, which may lead to short bowel syndrome or death.

Currently, there is no prenatal screening strategy for intestinal malrotation, and the feasibility and diagnostic performance of third-trimester obstetric ultrasound for detecting intestinal malrotation have never been formally evaluated.

Aim: To evaluate the diagnostic performance of third-trimester obstetric ultrasound in identifying the intestinal structures involved in high-risk intestinal malrotation associated with volvulus, using fetal MRI as the reference standard.

Methods : Eligible pregnant women will be identified during routine obstetric follow-up at Nîmes or Montpellier University Hospitals and enrolled exclusively in Montpellier. Each participant will undergo a third-trimester obstetric ultrasound and fetal MRI on the same day. Examinations will be performed independently by a senior obstetrician and a senior pediatric radiologist, both blinded to the other modality. Ultrasound visualization of mesenteric vessels, small bowel, and cecum will be compared with fetal MRI findings as the reference standard. Interobserver agreement for ultrasound interpretation will be assessed, and analyses will be stratified by gestational age. Participation duration is one day.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over the age of 18
* Good understanding of French
* Gestational age greater than or equal than 31 weeks
* Fetal MRI indication validated in multidisciplinary staff at weekly meetings of the Multidisciplinary Prenatal Diagnosis Center in Montpellier or Nimes
* Affiliation or beneficiary of a social security scheme
* Declaration of free and enlightened opposition

Exclusion Criteria:

* Complex fetal abdominal malformations responsible for difficult interpretation of imaging: heterotaxis with asplenia or polysplenium, diaphragmatic hernia, omphalocele, gastroschisis, digestive pathology, abdominal tumor, bladder exstrophy or megavessia.
* Fetal chromosomal abnormality
* Request for termination of pregnancy validated by a Multidisciplinary Pre-natal Diagnosis Center

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women with normal intestinal structure and requiring a fetal MRI for other reason
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Ultrasound localization of intestinal structure (mesenteric vessels, small bowel, gut) | At the visit 1 of the subjects
  The primary outcome will be ultrasound localization of intestinal structure (mesenteric vessels, small bowel, gut)

SECONDARY OUTCOMES:
normal meconium progression | At the visit 1 of the subjects
  Normal meconium progression will be described by the results of ultrasound examination and MRI

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malek MM, Burd RS. Surgical treatment of malrotation after infancy: a population-based study. J Pediatr Surg. 2005 Jan;40(1):285-9. doi: 10.1016/j.jpedsurg.2004.09.028. PMID 15868599
- [Background] Orzech N, Navarro OM, Langer JC. Is ultrasonography a good screening test for intestinal malrotation? J Pediatr Surg. 2006 May;41(5):1005-9. doi: 10.1016/j.jpedsurg.2005.12.070. PMID 16677901
- [Background] Dufour D, Delaet MH, Dassonville M, Cadranel S, Perlmutter N. Midgut malrotation, the reliability of sonographic diagnosis. Pediatr Radiol. 1992;22(1):21-3. doi: 10.1007/BF02011604. PMID 1594305
- [Background] Saguintaah M, Couture A, Veyrac C, Baud C, Quere MP. MRI of the fetal gastrointestinal tract. Pediatr Radiol. 2002 Jun;32(6):395-404. doi: 10.1007/s00247-001-0607-1. Epub 2002 Feb 16. PMID 12029338
- [Background] Boylan P, Parisi V. An overview of hydramnios. Semin Perinatol. 1986 Apr;10(2):136-41. PMID 3541223
- [Background] Veyrac C, Couture A, Saguintaah M, Baud C. [MRI of fetal GI tract]. J Gynecol Obstet Biol Reprod (Paris). 2005 Feb;34(1 Suppl):S14-7. doi: 10.1016/s0368-2315(05)82681-x. French. PMID 15767925
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Background] Veyrac C, Baud C, Prodhomme O, Saguintaah M, Couture A. US assessment of neonatal bowel (necrotizing enterocolitis excluded). Pediatr Radiol. 2012 Jan;42 Suppl 1:S107-14. doi: 10.1007/s00247-011-2173-5. Epub 2012 Mar 6. PMID 22395723
- [Background] Couture A, Veyrac C, Baud C, Saguintaahi M. [Imaging in neonatal intestinal obstruction]. JBR-BTR. 2005 Sep-Oct;88(5):259-61. No abstract available. French. PMID 16302344
- [Background] Veyrac C, Couture A, Saguintaah M, Baud C. MRI of fetal GI tract abnormalities. Abdom Imaging. 2004 Jul-Aug;29(4):411-20. doi: 10.1007/s00261-003-0147-2. Epub 2004 May 12. PMID 15136891
- [Background] Faure JM, Mousty E, Bigorre M, Wells C, Boulot P, Captier G, Fuchs F. Prenatal ultrasound diagnosis of cleft palate without cleft lip, the new ultrasound semiology. Prenat Diagn. 2020 Oct;40(11):1447-1458. doi: 10.1002/pd.5794. Epub 2020 Aug 17. PMID 32673416